CLINICAL TRIAL: NCT01259596
Title: A Randomized Controlled Trial (RCT)of Cognitive Behavioral Therapy-Telephone (CBT-T) for Late-Life Generalized Anxiety Disorder (GAD)
Brief Title: Telephone Psychotherapy for Late-Life Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010377; R01MH083664 (NIH)
Record Dates: First submitted 2010-11-12; First posted 2010-12-14 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: anxiety; rural; elderly
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (Active Comparator): Cognitive-behavioral therapy consists of psychoeducation, relaxation techniques, cognitive therapy, problem-solving, thought stopping, behavioral activation, exposure, coping with pain, sleep, and relapse prevention
  Interventions: Behavioral: cognitive behavioral therapy
- Nondirective supportive therapy (Active Comparator): Nondirective supportive therapy consists of providing a warm and accepting environment in which a person can reflect on their experiences, thoughts, and feelings
  Interventions: Behavioral: nondirective supportive therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — weekly individual psychotherapy by telephone for 12 weeks; 4 booster sessions
  Other Names: CBT
  Arms: Cognitive behavioral therapy
Behavioral: nondirective supportive therapy — weekly individual psychotherapy by telephone for 12 weeks; 4 booster sessions
  Other Names: NST
  Arms: Nondirective supportive therapy

SUMMARY:
The purpose of this study is to determine if cognitive-behavioral therapy (CBT)and supportive therapy delivered by telephone are effective for reducing worry and anxiety in rural older adults with Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
Older adults in rural locations often face significant barriers to treatment, including stigma, transportation, lack of local appropriately trained service providers, and impaired mobility. The proposed treatment is delivered in a workbook format and by telephone, which maximizes its portability. Treatment will be compared with nondirective supportive therapy, a very credible comparison condition equivalent to the intervention in therapist attention. We propose to randomize 88 adults ≥ 60 years with a diagnosis of GAD to either cognitive behavioral therapy delivered by telephone, or nondirective supportive therapy. The 2 primary treatment outcomes are anxiety symptoms as assessed by the Hamilton Anxiety Rating Scale, and worry symptoms as assessed by the Penn State Worry Questionnaire-Abbreviated. The proposed secondary outcomes are depressive symptoms, sleep, disability, and quality of life. Further, mediators and moderators of the treatment effect will also be examined. Mediators include process variables (therapeutic alliance, adherence, participant satisfaction, and treatment credibility) and new psychotropic medication use; moderators include demographic information (age, education, gender, race, income), psychiatric variables (baseline anxiety severity, baseline depressive disorders, baseline psychotropic medication use), medical comorbidity, and therapist assignment. Maintenance of response will be assessed over 6 months. This research has great public health significance, because it is a low-cost intervention with high potential for widespread dissemination, and it targets an underserved group - community-dwelling rural elders - who currently lack effective treatment interventions tailored to their needs.

ELIGIBILITY:
Inclusion Criteria:

* 60 years GAD Reside in rural county Proficient in English

Exclusion Criteria:

Current psychotherapy Active alcohol or substance abuse with use within last month Dementia or global cognitive impairment Psychotic symptoms Active suicidal ideation with plan and intent Change in psychotropic medications within last 1 month Significant hearing loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen A. Brenes, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenes GA, Danhauer SC, Lyles MF, Hogan PE, Miller ME. Telephone-Delivered Cognitive Behavioral Therapy and Telephone-Delivered Nondirective Supportive Therapy for Rural Older Adults With Generalized Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Oct;72(10):1012-20. doi: 10.1001/jamapsychiatry.2015.1154. PMID 26244854
- [Derived] Brenes GA, Danhauer SC, Lyles MF, Miller ME. Telephone-delivered psychotherapy for rural-dwelling older adults with generalized anxiety disorder: study protocol of a randomized controlled trial. BMC Psychiatry. 2014 Feb 8;14:34. doi: 10.1186/1471-244X-14-34. PMID 24506950

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive-behavioral Therapy: Cognitive-behavioral therapy consists of psychoeducation, relaxation techniques, cognitive therapy, problem-solving, thought stopping, behavioral activation, exposure, coping with pain, sleep, and relapse prevention
  psychotherapy: weekly individual psychotherapy by telephone for 12 weeks; 4 booster sessions
- Nondirective Supportive Therapy: Nondirective supportive therapy consists of providing a warm and accepting environment in which a person can reflect on their experiences, thoughts, and feelings
  psychotherapy: weekly individual psychotherapy by telephone for 12 weeks; 4 booster sessions
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Started | 70 | 71
Completed | 66 | 65
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 34 | 75
  >=65 years | 29 | 37 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 64 | 64 | 128
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 141

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Penn State Worry Questionnaire (PSWQ-A) at Week 13
Description: self-reported severity and frequency of worry the scores range from 8 to 40, with higher scores representing higher severity of worry. Higher scores represent worse outcome.
Time Frame: baseline to week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 65 | 64
units on a scale | -9.44 [-11.02 to -7.86] | -5.37 [-6.89 to -3.85]

2. Primary Outcome: Changes From Baseline in Hamilton Anxiety Rating Scale (HAM-A) at Week 13
Description: interviewer-rated severity of anxiety symptoms; the scores range from 0 to 56, with higher scores representing higher severity of anxiety. Higher scores represent worse outcome.
Time Frame: baseline to week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 64 | 64
units on a scale | -7.04 [-8.88 to -5.21] | -5.53 [-7.28 to -3.77]

3. Secondary Outcome: Changes From Baseline in Beck Depression Inventory (BDI) at 13 Weeks
Description: self report measure of depressive symptoms; scores range from 0 to 63, with a higher score representing higher levels of depressive symptoms Higher scores represent worse outcome.
Time Frame: baseline to week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 64 | 64
units on a scale | -10.77 [-12.73 to -8.81] | -7.54 [-9.44 to -5.64]

4. Secondary Outcome: Pepper Center Tool for Disability (PCT-D)
Description: self report measure of perceived difficulties with mobility and performing basic and advanced activities of daily living; the scale consists of 19 items; scores range from 19 to 114, with higher scores indicating more disability. Higher scores represent worse outcome.
Time Frame: week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 65 | 64
units on a scale | 1.71 [1.55 to 1.87] | 1.86 [1.70 to 2.01]

5. Secondary Outcome: Short Form (36) Health Survey (SF-36) to Week 13
Description: physical and emotional health related quality of life; The SF-36 is a self-report measure of health-related quality of life (HRQL) consisting of 36 items that form 8 subscales: physical functioning, role limitations due to physical health problems, role limitations due to emotional health problems, social functioning, freedom from pain, energy, emotional well-being, and general health perceptions. These 8 subscales are also combined into two domains: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). All of these scales range from 0 (maximum impairment) to 100 (no impairment). A lower score represents worse outcome.
Time Frame: week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 65 | 64
units on a scale | 60.5 [55.9 to 65.1] | 53.5 [49.1 to 57.9]

6. Secondary Outcome: Insomnia Severity Index (ISI)
Description: self-report symptoms of insomnia; scores range from 0 to 28 with higher scores indicating greater symptoms of sleep disturbance; higher score represents worse outcomes
Time Frame: week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 65 | 64
units on a scale | 8.70 [7.10 to 10.3] | 11.9 [10.4 to 13.4]

7. Secondary Outcome: Changes From Baseline in Generalized Anxiety Disorder-7 (GAD-7) to Week 13
Description: Diagnostic and Statistical Manual of Mental Disorders, IV edition (DSM-IV0) symptoms of Generalized Anxiety Disorder; scores range from 0 to 24 with higher scores indicating greater symptoms of GAD; higher score represents worse outcome
Time Frame: baseline to week 13
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Number analyzed (Participants) | 65 | 64
units on a scale | -5.63 [-6.82 to -4.44] | -3.27 [-4.40 to -2.14]

ADVERSE EVENTS:
Arm/Group | Cognitive-behavioral Therapy | Nondirective Supportive Therapy
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/71
Other Adverse Events (participants affected / at risk) | 4/70 | 4/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive-behavioral Therapy (N=70) | Nondirective Supportive Therapy (N=71)
serious adverse event (Psychiatric disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive-behavioral Therapy (N=70) | Nondirective Supportive Therapy (N=71)
adverse event (Psychiatric disorders) | 4 (4) | 4 (4) — 1SD increase in either PSWQ-A or BDI scores

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No